CLINICAL TRIAL: NCT01555138
Title: A Randomized, Double-blind, Parallel-group, 26-week Study Comparing the Efficacy and Safety of Indacaterol (Onbrez® Breezhaler® 150 mcg o.d.) With Salmeterol/Fluticasone Propionate (Seretide® Accuhaler® 50 mcg/500 mcg b.i.d.) in Patients With Moderate Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Indacaterol 150 mcg Once Daily (o.d.) With Salmeterol/Fluticasone Propionate 50 mcg/500 mcg Twice Daily (b.i.d.)
Acronym: INSTEAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2401; 2011-003732-31 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Indacaterol; Salmeterol/fluticasone propionate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 mcg once daily (o.d.) delivered via the Novartis single dose dry power inhaler (SDDPI) (Onbrez® Breezhaler®)
  Interventions: Drug: Indacaterol
- Salmeterol/fluticasone propionate (Active Comparator): Salmeterol 50 mcg /fluticasone propionate 500 mcg for inhalation delivered via a proprietary multi dose dry powder inhaler (MDDPI) device (Seretide® Accuhaler®) twice daily (b.i.d.)
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol is delivered via a SDDPI.
  Arms: Indacaterol
Drug: Salmeterol — Salmeterol/fluticasone is delivered via a MDDPI
  Arms: Salmeterol/fluticasone propionate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of indacaterol with salmeterol /fluticasone propionate treatment in patients with moderate chronic obstructive pulmonary disease who, on entry to the study are being treated with salmeterol /fluticasone propionate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate COPD (Stage II)
* Able to perform spirometry assessments
* Current or ex-smokers
* On treatment with the fixed-dose combination of salmeterol 50 µg/fluticasone propionate 500 µg MDDPI b.i.d. for the treatment of COPD for ≥ 3 months directly preceding Visit 1.

Exclusion Criteria:

* Having had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the past year.
* Having a history of, or current ECG abnormality
* Asthma

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (76):
- Argentina (17):
  - Novartis Investigative Site, Caba, Argentina
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, C A B A, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Villa María, Córdoba Province
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
- Colombia (3):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Italy (23):
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Cassano delle Murge, BA
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Forlì, FC
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Cassino, FR
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Sesto San Giovanni, Mi
  - Novartis Investigative Site, Cittadella, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Cuasso al Monte, VA
  - Novartis Investigative Site, Tradate, VA
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Verona, VR
- Malaysia (3):
  - Novartis Investigative Site, Wilayah Persekutuan, Kuala Lumpur
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Pulau Pinang
- Mexico (5):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Querétaro City, Querétaro
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
- Netherlands (3):
  - Novartis Investigative Site, Breda, Netherlands
  - Novartis Investigative Site, Helmond, Netherlands
  - Novartis Investigative Site, Rotterdam
- Spain (9):
  - Novartis Investigative Site, Loja, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Canet de Mar, Catalonia
  - Novartis Investigative Site, Corbera de Llobregat, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
- Switzerland (4):
  - Novartis Investigative Site, Muenchenstein, Switzerland
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Biel
  - Novartis Investigative Site, Gossau
- United Kingdom (9):
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle-upon-Tyne
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Hants, Southampton
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Chester
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Kettering
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, Surrey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Started | 293 | 288
Completed | 246 | 250
Not Completed | 47 | 38
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Abnormal Lab reults | 1 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 5 | 3
Not completed — Administrative problems | 8 | 0
Not completed — Withdrawal by Subject | 16 | 15
Not completed — Adverse Event | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate | Total
Number analyzed (Participants) | 293 | 288 | 581
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.39) | 66.8 (8.53) | 66.0 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 91 | 180
  Male | 204 | 197 | 401

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) at 12 Weeks (Imputed With LOCF): Treatment Comparisons
Description: Spirometry conducted to internationally accepted standards. Trough FEV1 defined as the mean of the FEV1 measurements at 23 h 10 min and 23 h 45 min post the Day 84 morning dose. The primary variable (imputed with last observation carried forward) will be analysed using a mixed model for the Per Protocol Set (PPS). The model will contain treatment as a fixed effect with the baseline FEV1 measurement, FEV1 prior to inhalation and FEV1 10-15 min post inhalation of salbutamol (components of reversibility at Visit 1) as covariates.
Time Frame: 12 weeks
Population: full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters | 1.591 (0.0276) | 1.604 (0.0281)

2. Secondary Outcome: Trough FEV1 (L) at Week 26 (Imputed With LOCF): Treatment Comparisons
Description: Trough FEV1 is defined as the average of the 23 h 10 min and the 23 h 45 min values taken in the clinic at Visit 11.
Time Frame: 26 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters | 1.567 (0.0302) | 1.569 (0.0307)

3. Secondary Outcome: FEV1 (L) at Individual Time Points After 12 Weeks Treatment: Treatment Comparisons
Description: FEV1 at each time point, for each visit, will be analyzed using the same mixed model as specified for the primary analysis. Least squares means will be displayed by treatment group.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters
  -50 min pre-dose | 1.601 (0.0281) | 1.588 (0.0286)
  30 min post-dose, | 1.667 (0.0207) | 1.656 (0.0208)
  1h post-dose, | 1.693 (0.0285) | 1.684 (0.0293)
  2h post-dose | 1.705 (0.0291) | 1.708 (0.0300)
  4h post-dose | 1.670 (0.0215) | 1.699 (0.0216)
  23h 10 min post-dose | 1.577 (0.0277) | 1.591 (0.0284)
  23h 45 min post-dose | 1.597 (0.0283) | 1.613 (0.0291)
  -15 min pre-dose | 1.623 (0.0282) | 1.616 (0.287)
  5 min post-dose | 1.631 (0.0209) | 1.613 (0.0209)

4. Secondary Outcome: FEV1 (L) at Individual Time Points After 26 Weeks Treatment: Treatment Comparisons
Description: FEV1 at each time point, for each visit, will be analyzed using the same mixed model as specified for the primary analysis. Least squares means will be displayed by treatment group .
Time Frame: 26 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters
  -50 min pre-dose | 1.569 (0.0301) | 1.582 (0.0304)
  30 min post-dose, | 1.670 (0.0244) | 1.656 (0.0244)
  1h post-dose, | 1.676 (0.0317) | 1.677 (0.0324)
  2h post-dose | 1.700 (0.0318) | 1.693 (0.0325)
  4h post-dose | 1.664 (0.0320) | 1.663 (0.0328)
  23h 10 min post-dose | 1.551 (0.0305) | 1.559 (0.0310)
  23h 45 min post-dose | 1.574 (0.313) | 1.575 (0.0318)
  -15 min pre-dose | 1.576 (0.0294) | 1.595 (0.0300)
  5 min post-dose | 1.630 (0.0304) | 1.630 (0.0310)

5. Secondary Outcome: FVC Over 26 Weeks of Treatment
Description: FVC at each time point, for each visit, will be analyzed using the same mixed model as specified for the primary analysis. Least squares means will be displayed by treatment group.
Time Frame: 12 and 26 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters
  12 weeks | 3.090 (0.0457) | 3.064 (0.0466)
  26 weeks | 3.057 (0.0512) | 3.062 (0.0520)

6. Secondary Outcome: Analysis of AUC (5 Min - 4 h) for FEV1 (L) at Week 12 and Week 26: Treatment Comparison
Description: The standardized (with respect to the length of time) AUC for FEV1 will be calculated between 5 min and 4 h post morning dose as the sum of trapezoids divided by the length of time at Day 84 (Visit 6) and Day 182 (Visit 10). Scheduled (not actual) time points are to be used. FEV1 measurements taken within 6 h of rescue use will be set to missing before the standardized AUC is calculated.
Time Frame: 12 and 26 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Liters
  Week 12 | 1.689 (0.0201) | 1.689 (0.0203)
  Week 26 | 1.683 (0.0304) | 1.682 (0.0310)

7. Secondary Outcome: TDI Focal Score at Week 12 and Week 26: Treatment Comparisons
Description: The Transition Dyspnea Index (TDI) total score after 12 and 26 weeks of treatment will be analyzed using the same mixed model as specified for the primary analysis with the Baseline Dyspnea Index (BDI) total score as the baseline.Total score ranging - 9 to + 9. The lower the score, the more deterioration in severity of dyspnea. One additional option in each category, which does not contribute to the score, allows for circumstances in which impairment is due to reasons other than dyspnea.
Time Frame: 12 and 26 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
Units on a scale
  12 weeks | 1.89 (0.499) | 1.69 (0.509)
  26 weeks | 2.58 (0.543) | 2.70 (0.552)

8. Secondary Outcome: Number of COPD Exacerbations Per Patient Over 26 Weeks: Treatment Comparisons (Without Imputation; Full Analysis Set)
Description: The number of exacerbations during the 26 week treatment period will be analyzed using a generalized linear model assuming a negative binomial distribution.
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
participants
  none | 233 | 215
  one | 47 | 57
  two | 11 | 15
  three | 2 | 1
  Greater than or equal to four | 0 | 0

9. Secondary Outcome: Mean Daily Number of Puffs of Rescue Medication Used Over 26 Weeks of Treatment
Description: The mean daily number of puffs of rescue medication taken by the patient will be derived. If the number of puffs is missing for part of the day (either morning or evening) then a half day will be used in the denominator. Rescue medication data recorded during the 14 day run-in period will be used to calculate the baseline. The mean change from baseline in the daily number of puffs of rescue medication will be analyzed using the same mixed model as specified for the primary analysis, with the baseline FEV1 replaced with the baseline daily rescue use.
Time Frame: 12 and 26 weeks
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
number of puffs
  Baseline | 1.82 (2.274) | 1.83 (2.035)
  Week 12 | 1.50 (1.883) | 1.45 (1.697)
  Week 26 | 1.37 (1.775) | 1.37 (1.678)

10. Secondary Outcome: Rescue Medication Use Over 26 Weeks: Percentage of 'Days With no Rescue Use'
Description: A 'day with no rescue use' is defined from diary data as any day where the patient has taken no puffs of rescue medication. The percentage of 'days with no rescue use' will be derived and analyzed as for the percentage of 'nights with no nighttime awakenings'.
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: % of Days
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
% of Days | 52.8 (3.71) | 54.6 (3.68)

11. Secondary Outcome: St Georges Respiratory Questionnaire for COPD
Description: A Total and three component scores are calculated: Symptoms; Activity; Impacts. Each component of the questionnaire is scored separately:The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the result as a percentage: Score = 100 x Summed weights from all positive items in that component divided by Sum of weights for all items in that component The Total score is calculated in similar way: Score = 100 x Summed weights from all positive items in the questionnaire divided by Sum of weights for all items in the questionnaire Sum of maximum possible weights for each component and Total: Symptoms 566.2 Activity 982.9 Impacts 1652.8 Total (sum of maximum for all three components) 3201.9 The proportion of patients who achieve a clinically important improvement of at least 4 units in the total SGRQ will be analyzed. The higher the score the more symptoms of disease are present.
Time Frame: 12 and 26 weeks
Population: Full Analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Indacaterol | Salmeterol/Fluticasone Propionate
Number analyzed (Participants) | 293 | 288
scores on a scale
  Week 12 | 32.8 (1.58) | 32.9 (1.61)
  Week 26 | 33.1 (1.87) | 33.5 (1.93)

ADVERSE EVENTS:
Groups:
- Indacaterol: Indacaterol 150 μg once daily (o.d.) delivered via the Novartis single dose dry power inhaler (SDDPI) (Onbrez® Breezhaler®)
- Salmeterol/Fluticasone: Salmeterol 50 μg /fluticasone propionate 500 μg for inhalation delivered via a proprietary multi dose dry powder inhaler (MDDPI) device (Seretide® Accuhaler®) twice daily (b.i.d.)
Arm/Group | Indacaterol | Salmeterol/Fluticasone
Serious Adverse Events (participants affected / at risk) | 5/293 | 17/288
Other Adverse Events (participants affected / at risk) | 70/293 | 85/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=293) | Salmeterol/Fluticasone (N=288)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=293) | Salmeterol/Fluticasone (N=288)
Nasopharyngitis (Infections and infestations) | 15 | 18
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 60 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial